CLINICAL TRIAL: NCT04966988
Title: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Brief Title: Multimodal Imaging Evaluation and Prognostic Analysis of Cardiac Allograft Vasculopathy in Heart Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Xie Mingxing (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai Zhongshan Hospital (Other); Henan Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xie Mingxing, MD, PhD,FACC, FAHA, FASE, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2021 V 1.0
Record Dates: First submitted 2021-07-10; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CAV 0(Not significant): No detectable angiographic lesion
- CAV 1 (Mild): Angiographic left main (LM) <50%, or primary vessel with maximum lesion of <70%, or any branch stenosis <70% (including diffuse narrowing) without allograft dysfunction
- CAV 2 (Moderate): Angiographic LM <50%; a single primary vessel≥70%, or isolated branch stenosis ≥70% in branches
- CAV 3 (Severe): Angiographic LM≥50%, or two or more primary vessels ≥70% stenosis, or isolated branch stenosis≥70%in all 3 systems; or CAV1 or CAV2 with allograft dysfunction (defined as LVEF≤45% usually in the presence of regional wall motion abnormalities) or evidence of significant restrictive physiology

SUMMARY:
The aim is to (1) establish a system of multimodal imaging technology; (2) jointly apply multimodal imaging technology to diagnose of cardiac allograft vasculopathy of heart transplantation; (3) construct a multimodal imaging technology prediction model of adverse events, screening the best non-invasive imaging prediction indicators.

DETAILED DESCRIPTION:
This study will enrolled 1000 HT patients, and the cardiac allograft vasculopathy will be evaluated by multimodal imaging technology. The aim is to (1) establish a system of multimodal imaging technology; (2) jointly apply multimodal imaging technology to diagnose of cardiac allograft vasculopathy of heart transplantation; (3) construct a multimodal imaging technology prediction model of adverse events, screening the best non-invasive imaging prediction indicators.

ELIGIBILITY:
Inclusion Criteria:

• Heart transplantation after January 1st, 2015.

Exclusion Criteria:

•Age < 18 years at the time of transplantation; Died within 48 h; Heart-lung transplantation; Heart/kidney transplantation; Re-transplanted within 7 days after transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult HT recipients were consecutive prospectively enrolled who underwent transthoracic echocardiography for surveillance at their routine follow-up
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
All cause death | up to 10 year
  All cause death after HT was obtained via telephone interview with family members; contact with his/her physicians; or hospital records

SECONDARY OUTCOMES:
Major adverse cardiac events | 5 year and 10 year
  Major adverse cardiac events after the inclusion of the study was obtained via telephone interview with family members; contact with his/her physicians; or hospital records

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PhD, Principal Investigator — Department of Ultrasound, Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No